CLINICAL TRIAL: NCT03869047
Title: Dexmedetomidine Added to Bupivacaine Versus Bupivacaine inTransincisionalU/S Guided Quadratus Lumborum Block in Open Renal Surgeries , A New Technique :Prospective, Randomized Double- Blinded Study
Brief Title: Dexmedetomidine Added to Bupivacaine Versus Bupivacaine inTransincisionalU/S Guided Quadratus Lumborum Block in Open Renal Surgeries , A New Technique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 14/2019
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quadratus lumborum block(dexmedetomidine+bupivacaine) (Active Comparator): patients will receive combined general anesthesia and Quadratuslumborum block( transincisional ie before wound closure)with 19 mL of bupivacaine 0.20%plus 1 mic/kg of dexmedetomidine ,total volume 20 ml.
  Interventions: Drug: Dexmedetomidine +bupivacaine
- quadratus lumborum block(bupivacaine) (Active Comparator): patients will receive combined general anesthesia and quadratus lumborum block (transincisional) with 20 ml of bupivacaine 0.20%.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine +bupivacaine — patients will receive combined general anesthesia and Quadratuslumborum block( transincisional ie before wound closure)with 19 mL of bupivacaine 0.20%plus 1 mic/kg of dexmedetomidine, total volume 20 ml
  Arms: quadratus lumborum block(dexmedetomidine+bupivacaine)
Drug: Bupivacaine — patients will receive combined general anesthesia and quadratus lumborum block (transincisional) with 20 ml of bupivacaine 0.20% .
  Arms: quadratus lumborum block(bupivacaine)

SUMMARY:
The purpose of this study is to compare the addition of dexmedetomidine to bupivacaine versus bupivacaine only in anterior QLblock(transincisional) , where the local anesthetic will be applied before wound closure at the end of surgery through the wound . in combination with general anesthesia in elective open renal surgery with regard to Postoperative pain control,hemodynamic stability, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* physical status American Society of Anesthesiologist (ASA) I or II

Exclusion Criteria:

* Patients refusal
* A body mass index (BMI) >30 kg/m2
* ASA physical status >II
* major illnesses (e.g., cardiac, respiratory, renal, hepatic or neurological)
* Coagulation abnormalities
* Infection at the injection site
* Allergy or contraindications to the drugs used in the study
* History of drug addiction or alcohol abuse
* A psychiatric illness, or mental retardation interfering with the evaluation of pain scores or PCA programs .

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | 1st 24 hour postoperatively
  After extubation, an intravenous patient - controlled system, will be connected to the patient (Accufuser plus 100 ml) will be prepared with 60 ml isotonic saline containing 60 mg morphine , it will be programmed to give 0.5 ml bolus dose with lockout interval of 8 minutes. Time to first bolus will be recorded considering extubation time is the zero time

SECONDARY OUTCOMES:
the secondary outcomes will be the total opioid consumption postoperatively | 1st 24 hour
  PCA will prepared with 60 mL of normal saline containing 60 mg of morphine, and the system will be programmed to give a 0.5 mL bolus dose with a lockout interval of 8 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes